CLINICAL TRIAL: NCT05568199
Title: Udall Project 1 Aim 4
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007781
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Parkinsons Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients will make one visit to the M Health Clinical Research Unit (CRU) after overnight withdrawal of PD medications (still on-DBS) and undergo motor and cognitive assessments in the following three conditions:
  1. clinically-optimized stimulation
  2. model-based stimulation directed towards motor subregions of STN and GPi
  3. model-based stimulation directed towards associative/limbic subregions of STN/GPi
  Randomized to start with condition1 assessment
- Group 2: Patients will make one visit to the M Health Clinical Research Unit (CRU) after overnight withdrawal of PD medications (still on-DBS) and undergo motor and cognitive assessments in the following three conditions:
  1. clinically-optimized stimulation
  2. model-based stimulation directed towards motor subregions of STN and GPi
  3. model-based stimulation directed towards associative/limbic subregions of STN/GPi
  Randomized to start with condition 2 assessment
- Group 3: Patients will make one visit to the M Health Clinical Research Unit (CRU) after overnight withdrawal of PD medications (still on-DBS) and undergo motor and cognitive assessments in the following three conditions:
  1. clinically-optimized stimulation
  2. model-based stimulation directed towards motor subregions of STN and GPi
  3. model-based stimulation directed towards associative/limbic subregions of STN/GPi
  Randomized to start with condition 3 assessment

SUMMARY:
By defining the strength and direction of connectivity patterns at rest and during movement across the basal ganglia-thalamocortical (BGTC) network we will characterize the role of individual circuits in motor performance and cognitive function, paving the way for future development of optimization algorithms for DBS that take advantage of this understanding.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a DBS system
* Existing 7T imagery (either done as standard-of-care or done as part of Noam Harel's study, IRB #1210M22183)
* Diagnosed with idiopathic Parkinson's Disease
* Minimum age 21 years

Exclusion Criteria:

* Other significant neurological disorder, as determined by PI
* Diagnosis of dementia
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants are identified by clinicians and trained research personnel through the movement disorder clinic. Patients are identified during the University of Minnesota DBS surgery candidacy evaluation process.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Motor association with pathway activation patterns | 6 months post surgery
  associate pathway activation patterns with motor (UPDRS-III) outcome obtained during standard of care and research appointments.
Cognitive outcome 1 association with pathway activation pattern | 6 months post surgery
  associate pathway activation patterns with cognitive outcome obtained during standard of care and research appointments.
  One primary cognitive outcome measure will be the D-KEFS Letter Fluency test. Another primary cognitive measure will be the Stroop Color Word total score. Secondary measures will include the Beck Depression Inventory (BDI)-II and Apathy Scale total scores.
Cognitive outcome 2 association with pathway activation pattern | 6 months post surgery
  associate pathway activation patterns with cognitive outcome obtained during standard of care and research appointments.
  cognitive measure will be the Stroop Color Word total score.
Cognitive outcome 3 association with pathway activation pattern | 6 months post surgery
  associate pathway activation patterns with cognitive outcome obtained during standard of care and research appointments.
  cognitive measure will include the Beck Depression Inventory (BDI)-II
Cognitive outcome 4 association with pathway activation pattern | 6 months post surgery
  associate pathway activation patterns with cognitive outcome obtained during standard of care and research appointments.
  cognitive measure will include the Apathy Scale total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Vitek, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University Of Minnesota, Minneapolis, Minnesota, United States